CLINICAL TRIAL: NCT02856854
Title: A Phase 1b, Randomized, Double-Blinded, Multiple-Dose, Placebo Controlled, Crossover Study To Evaluate The Safety, Tolerability And Pharmacokinetic Effects Of A Metyrapone And Oxazepam Combination (EMB-001) When Co-Administered With Cocaine
Brief Title: A Study of Metyrapone and Oxazepam Combination Product (EMB-001) and Cocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ERL-002; U01DA038879 (NIH)
Record Dates: First submitted 2016-07-22; First posted 2016-08-05 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Metyrapone; Oxazepam; Cocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMB-001 (oral) (Experimental): EMB-001 will be orally administered for 7 consecutive days, twice daily for 6 days followed on the last day by one EMB-001 oral dose (QD) in the morning. Three hours later Cocaine IV or Saline IV will be administered followed 2 hours by the other (saline or cocaine).
  Interventions: Drug: EMB-001; Drug: Cocaine IV; Drug: Saline IV
- Placebo (oral) (Placebo Comparator): PLB-to-match EMB-001 will be orally administered for 7 consecutive days, BID for 6 days, followed on the last day by one PLB oral dose in the morning. Three hours later Cocaine IV or Saline IV will be administered followed 2 hours by the other (saline or cocaine).
  Interventions: Drug: Placebo; Drug: Cocaine IV; Drug: Saline IV

INTERVENTIONS:
Drug: EMB-001 — EMB-001 is a combination of metyrapone (720mg per dose in this study) and oxazepam (24mg per dose in this study)
  Other Names: metyrapone and oxazepam
  Arms: EMB-001 (oral)
Drug: Placebo — EMB-001 matched placebo
  Other Names: oral placebo
  Arms: Placebo (oral)
Drug: Cocaine IV — Cocaine administered at doses of 20 and 40mg
  Other Names: IV cocaine
Drug: Saline IV — Cocaine matched placebo
  Other Names: IV saline

SUMMARY:
EMB-001 is a combination of 2 drugs: the cortisol synthesis inhibitor, metyrapone (Metopirone®), and the benzodiazepine receptor agonist, oxazepam (original trade name Serax®; now marketed as oxazepam (generic) only).

This Phase 1b cocaine interaction study is being conducted in order to assess the safety and PK of EMB-001 and cocaine in combination.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blinded, multiple-dose, PLB controlled, 2-period, 4-sequence, crossover study design.

After establishing eligibility approximately 16 subjects with cocaine use disorder will be randomized to one of four sequences.

Treatment periods will be separated by a 7-day in-patient washout period. EMB-001/PLB will be orally administered for 7 consecutive days, BID for 6 days (starting on Day 1 and Day 15) followed on the last day (Day 7 and Day 21) by one EMB-001/PLB oral dose in the morning. Infusion of 40 mg IV cocaine and IV saline-to-match cocaine infusion will be administered in a randomized order, 2 hours apart, starting 3 hours after the last morning EMB-001/PLB oral administration.

The subjects will be discharged from the research clinic 2 days after the last dose of cocaine, and will have a follow-up visit 7 days after last dose.

ELIGIBILITY:
Inclusion Criteria:

* non-treatment-seeking cocaine users with a positive urine toxicology screen for cocaine at least once during screening
* have a medical history and physical examination that demonstrate no clinically significant contraindication for participating in the study
* males must use contraception; females must be of non-childbearing potential

Exclusion Criteria:

* drug allergies or reactions to metyrapone or benzodiazepines, or severe hypersensitivity reactions (like angioedema) to any drugs
* history of clinically significant adverse reaction to cocaine
* a low out-of-range serum cortisol value at screening or subjects who have a heightened likelihood of having adrenal insufficiency, or have signs or a history of adrenal insufficiency or confounders of the levels of cortisol and/or cortisol binding globulin
* treatment with glucocorticoids
* history of seizures, benzodiazepine use disorder, respiratory disease, neurologic or neuromuscular disease, liver disease or cardiovascular disease
* other psychiatric or substance use disorders of clinical significance, or suicidality
* clinically significant finding on medical history, physical examination, clinical laboratory tests, vital signs or ECGs
* use of any other drugs
* abnormal BP or HR
* positive urine drug screen at for alcohol or any drug other than marijuana (THC) or cocaine
* positive serology test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Antibody (HCVAb)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-17 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 29 Days
  Adverse event data (including clinically significant changes in laboratory values) will be compiled for EMB-001 and placebo cohorts.
Vital signs | 29 days
  Blood Pressure (BP) and heart rate (HR) measures during saline infusions will be compared to HR and BP after cocaine infusion (40 mg). Changes in BP and HR induced by cocaine infusion along with EMB-001 will be compared to those with EMB-001-matched placebo.
ECGs | 29 days
  Changes in ECG readings during saline infusion will be compared to those taken during cocaine infusion along with EMB-001 will be compared to those with EMB-001-matched placebo.

SECONDARY OUTCOMES:
PK Parameter EMB-001 | 21 days
  Cmax (maximum concentration) of EMB-001 will be compared when taken alone and when taken with cocaine
PK Parameter Cocaine | 21 days
  Cmax (maximum concentration) of cocaine will be compared when taken alone and when taken with EMB-001
PK Parameter EMB-001 | 21 days
  AUC (area under the curve) of EMB-001 will be compared when taken alone and when taken with cocaine
PK Parameter Cocaine | 21 days
  AUC (area under the curve) of Cocaine will be compared when taken alone and when taken with EMB-001

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince & Associates
Locations (1):
- Vince & Associates, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Every three months, the NIDA DSMB will convene to review the overall safety data, as well as data on safety summarized by treatment condition. As per NIH guidelines, the objective of these reviews will be to determine whether continued conduct of the trial poses any undue risk for participants. Blinded data tables, figures and/or listings will be provided to the Data Safety Monitoring Board (DSMB).
Supporting Information: Study Protocol, CSR
Time Frame: Every three months- blinded results
Access Criteria: A DSMB report is prepared an submitted via NIDA.

REFERENCES:
- [Background] Kablinger AS, Lindner MA, Casso S, Hefti F, DeMuth G, Fox BS, McNair LA, McCarthy BG, Goeders NE. Effects of the combination of metyrapone and oxazepam on cocaine craving and cocaine taking: a double-blind, randomized, placebo-controlled pilot study. J Psychopharmacol. 2012 Jul;26(7):973-81. doi: 10.1177/0269881111430745. Epub 2012 Jan 11. PMID 22236504